CLINICAL TRIAL: NCT06702813
Title: Physiological Effects and Safety of Continuous High-frequency Oscillatory Ventilation in ICU Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSZZ202411
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Atelectasis, Postoperative; Hypoxia; Critical Illness
Keywords: HFOV; EIT; atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis; Hypoxia; Critical Illness

STUDY DESIGN:
Intervention Model Description: Interventional study evaluating the beneficial impact of continuous high frequency oscillatory ventilation in ICU patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHFO group (Experimental): After checking the availability of the CHFO machine (MetaNeb® system), the inclusion and non-inclusion criteria, the patient is included. The following procedures are performed:
  1. installation of an EIT belt in the 4th or 5th intercostal space (Pulmovista® 500, Dräger);
  2. continuous recording of digital and analogic data after collecting initial data from the patient within 10 minutes before CHFO treatment, successive 10-minutes CHFO were performed. At the end of the treatment, all the data is collected.
  Interventions: Device: High-Frequency Oscillatory Ventilation

INTERVENTIONS:
Device: High-Frequency Oscillatory Ventilation — Administer 10 minutes of high-frequency oscillatory ventilation in awake ICU patients.

SUMMARY:
Atelectasis, hypoxemia, and ineffective sputum clearance are common problems in ICU patients. Continuous High-Frequency Oscillation (CHFO) is often considered to have a protective effect on the lungs. CHFO provides effective gas exchange at supraphysiological frequencies while minimizing pressure fluctuations, producing tidal volumes smaller than dead space, and adjusting around a continuously expanding pressure to optimize end-expiratory lung volume (EELV), thereby improving lung function by achieving and maintaining lung recruitment. However, the physiological effects and safety of CHFO in awake critically ill patients are still lacking relevant research. The objective of this study is to evaluate the comfort, safety, and efficacy of CHFO in awake critically ill patients.

DETAILED DESCRIPTION:
This is an interventional study evaluating the beneficial impact of CHFO (Continuous High Frequency Oscillatory Ventilation) in awake ICU patients with atelectasis on ventilatory function.

This therapeutic study aims to treat patients using the CHFO machine (MetaNeb system). The study involves comparing pulmonary pathophysiological parameters before and after CHFO treatment in awake patients with atelectasis.

The primary outcome is the difference in chest electrical impedance tomography (EIT) measurements taken at the end of CHFO treatment (10 minutes) compared to the baseline value measured at the beginning of the protocol.

The minimum number of subjects to enroll in this study is 45 patients. Intermediate analyses are planned after every 5 patients to reassess the required number of patients.

Baseline data collected at the beginning of the protocol include pulse oximetry and measurements of heart rate and blood pressure. During the treatment, pulse oximetry and measurements of heart rate and blood pressure will be collected. At the end of the treatment, arterial blood gas analysis, heart rate, and blood pressure will be measured. EIT data will be collected at 10 minutes before the start of CHFO, during treatment, and 10 minutes after the treatment. At the end of the treatment, collect patients' subjective ratings of treatment comfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 and younger than 90 years;
* Admitted to the ICU after December 1, 2024, who are alert, with a GCS of 15, normal comprehension, and able to communicate clearly through speech or writing.
* Patients with atelectasis, who are receiving oxygen therapy, high-flow oxygen, or are on a ventilator via tracheostomy.
* Signed informed consent for MetaNeb treatment.

Exclusion Criteria:

* Refusal to participate in the proposed study.
* Age < 10 years;
* Pregnancy;
* Significant hemodynamic instability defined as an increase of more than 20% in catecholamine doses in the last hour, despite optimization of blood volume, for a target mean blood pressure between 65 and 75 mmHg.
* Participation in another trial within 30 days prior to meeting eligibility criteria;
* Severe chronic respiratory disease requiring long-term oxygen therapy or home mechanical ventilation;
* Pneumothorax. With a clear tracheoesophageal fistula

Ages: 18 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-11-19 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
EIT | Baseline, during the treatment, and at the end of the intervention (10th minute).
  In EIT monitoring, a 16-electrode belt was placed around the chest to record signals. Measurements will be taken at three time points: (1) within 10 minutes before the start of CHFO, (2) during the treatment, and (3) within 10 minutes after its completion.

SECONDARY OUTCOMES:
SpO2 before, during and after the CHOF treatment | Baseline, during the treatment, and at the end of the intervention (10th minute).
  The SpO2 will be measured. Measurements will be taken at three time points: (1) Within 10 minutes before the start of CHFO and (2) During the treatment, and (3)within 10 minutes after its completion.
Mean arterial pressure | Baseline, during the treatment, and at the end of the intervention (10th minute).
  Mean arterial pressure will be measured. Measurements will be taken at three time points: (1) Within 10 minutes before the start of CHFO and (2) During the treatment, and (3)within 10 minutes after its completion.
Comfort Rating | Within 10 minutes after the treatment
  To have patients rate their comfort level with the treatment using the Numeric Rating Scale (NRS) after the treatment is completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China